CLINICAL TRIAL: NCT02713126
Title: Inorganic Nitrite to Enhance Benefits From Exercise Training in Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Inorganic Nitrite to Amplify the Benefits and Tolerability of Exercise Training in Heart Failure With Preserved Ejection Fraction (HFpEF) (INABLE-Training)
Acronym: INABLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barry Borlaug (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Barry Borlaug, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-001467; R01HL128526 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Nitrite; Nitrites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will undergo cardiac exercise training and receive inhaled or oral placebo three times per day for 12 weeks while wearing an accelerometer
  Interventions: Drug: Placebo; Device: Accelerometer; Other: Cardiac Exercise Training
- Sodium Nitrite (Active Comparator): Subjects will undergo cardiac exercise training and receive inhaled or oral sodium nitrite three times per day for 12 weeks while wearing an accelerometer
  Interventions: Drug: Sodium Nitrite; Device: Accelerometer; Other: Cardiac Exercise Training

INTERVENTIONS:
Drug: Placebo — administered orally or inhaled, taken every 4 hours or 3 times per day during waking hours for 12 weeks
  Arms: Placebo
Drug: Sodium Nitrite — administered orally or inhaled, 40 mg, taken every 4 hours or 3 times per day during waking hours for 12 weeks
  Other Names: Nitrite
  Arms: Sodium Nitrite
Device: Accelerometer — External triaxial accelerometer is worn externally at the hip during exercise training sessions, and day/night to continuously measure activity levels, removed for bathing only.
Other: Cardiac Exercise Training — Cardiac rehabilitation exercise training consisting of supervised endurance and strength exercise training of approximately one hour, 3 times per week for 12 weeks.

SUMMARY:
Participants with heart failure with preserved ejection fraction will undergo 12 weeks of cardiac rehabilitation for exercise training (ET) and be randomized to either sodium nitrite or placebo through the training period. Study drug is administered 3 times daily with one of these doses being 30 minutes prior to onset of ET sessions throughout the12 week trial. The objective is to determine if the sodium nitrite improves the clinical responses and tolerability of ET.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Symptoms of dyspnea (II-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
* Ejection Fraction (EF) of > or = 50% determined on most recent imaging study within the preceding 5 years, with no change in clinical status suggesting potential for deterioration in systolic function
* One of the following:

  * Previous hospitalization for Heart Failure (HF) with radiographic evidence (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) of pulmonary congestion or
  * Catheterization documented elevated filling pressures at rest (Pulmonary Capillary Wedge Pressure (PCWP)= ≥15 or Left Ventricular End-Diastolic Pressure (LVEDP) ≥18) or with exercise (PCWP ≥25) or
  * Elevated Natruretic Peptide-proBNP (>400 pg/ml) or B-Type Natriuretic Peptide (BNP)(>200 pg/ml) or
  * Echo evidence of diastolic dysfunction/elevated filling pressures manifest by medial E/e' ratio≥15 and/or left atrial enlargement and chronic treatment with a diuretic for signs or symptoms of heart failure
* Heart failure is primary factor limiting activity as indicated by answering # 2 to the following question:

My ability to be active is most limited by:

1. Joint, foot, leg, hip or back pain
2. Shortness of breath and/or fatigue and/or chest pain
3. Unsteadiness or dizziness
4. Lifestyle, weather, or I just don't like to be active

   * No chronic nitrate therapy or not using intermittent sublingual nitroglycerin (requirement for >1 sublingual nitroglycerin per week).
   * No daily use of phosphodiesterase 5 (PDE5) inhibitors or soluble guanylyl cyclase activators and willing to withhold as needed use of PDE5 inhibitors for duration of study
   * Ambulatory (not wheelchair / scooter dependent)
   * Body size allows wearing of the accelerometer belt as confirmed by ability to comfortably fasten the test belt provided for the screening process.
   * Willingness to wear the accelerometer belt for the duration of the trial

Exclusion Criteria:

* Recent (< 1 month) hospitalization for heart failure
* Ongoing requirement for PDE5 inhibitor, organic nitrate or soluble guanylyl cyclase activators
* Hemoglobin (Hgb) < 8.0 g/dl within 30 days prior to randomization
* Glomerular Filtration Rate (GFR) < 20 ml/min/1.73 m2 within 30 days prior to randomization
* Systolic blood pressure < 115 mmHg seated or < 90 mmHg standing
* Resting Heart Rate > 110
* Previous adverse reaction to the study drug which necessitated withdrawal of therapy
* Significant chronic obstructive pulmonary disease that is a primary contributor to symptoms, in the opinion of the Investigator.
* Ischemia thought to contribute to dyspnea, in the opinion of the Investigator.
* Documentation of previous Ejection Fraction < 40%
* Acute coronary syndrome within 3 months defined by electrocardiographic (ECG) changes and biomarkers of myocardial necrosis (e.g., troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
* Percutaneous Coronary Intervention, coronary artery bypass grafting, or new biventricular pacing within past 3 months
* Obstructive hypertrophic cardiomyopathy
* Known infiltrative cardiomyopathy (amyloid)
* Constrictive pericarditis or tamponade
* Active myocarditis
* Complex congenital heart disease
* Active collagen vascular disease
* More than mild aortic or mitral stenosis
* Intrinsic (prolapse, rheumatic) valve disease with more than moderate mitral, tricuspid or aortic regurgitation
* Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, International Normalized Ratio (INR) > 1.7 in the absence of anticoagulation treatment
* Terminal illness (other than HF) with expected survival of less than 1 year
* Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months.
* Inability to comply with planned study procedures
* Pregnancy or breastfeeding mothers

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-09; Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borlaug BA, Koepp KE, Reddy YNV, Obokata M, Sorimachi H, Freund M, Haberman D, Sweere K, Weber KL, Overholt EA, Safe BA, Omote K, Omar M, Popovic D, Acker NG, Gladwin MT, Olson TP, Carter RE. Inorganic Nitrite to Amplify the Benefits and Tolerability of Exercise Training in Heart Failure With Preserved Ejection Fraction: The INABLE-Training Trial. Mayo Clin Proc. 2024 Feb;99(2):206-217. doi: 10.1016/j.mayocp.2023.08.031. Epub 2023 Dec 21. PMID 38127015
- [Derived] Alogna A, Koepp KE, Sabbah M, Espindola Netto JM, Jensen MD, Kirkland JL, Lam CSP, Obokata M, Petrie MC, Ridker PM, Sorimachi H, Tchkonia T, Voors A, Redfield MM, Borlaug BA. Interleukin-6 in Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2023 Nov;11(11):1549-1561. doi: 10.1016/j.jchf.2023.06.031. Epub 2023 Aug 9. PMID 37565977
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Sodium Nitrite
Started | 36 | 56
Completed | 36 | 37
Not Completed | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sodium Nitrite | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73.5 [68.7 to 76.5] | 72.0 [64.9 to 76.0] | 72.4 [66.4 to 76.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 16 | 23 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 35 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Rate of Oxygen (VO2)
Description: Exercise capacity as measured by the peak rate of oxygen (VO2) consumption achieved during exercising testing. Peak VO2 is expressed as milliliters of oxygen per kilogram of body mass per minute.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Placebo | Sodium Nitrite
Number analyzed (Participants) | 34 | 31
ml/min/kg | 0.85 (2.10) | 0.70 (1.51)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite; Test type: Superiority; p = 0.770, t-test, 2 sided

2. Secondary Outcome: Change in Daily Activity Levels
Description: The change in daily activity levels as assessed by accelerometer data and reported as average accelerometry units.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: accelerometry units (AU)
Arm/Group | Placebo | Sodium Nitrite
Number analyzed (Participants) | 27 | 22
accelerometry units (AU) | -4 (51) | 23 (70)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite; Test type: Superiority; p = 0.087, t-test, 2 sided

3. Secondary Outcome: Change in Cardiac Hemodynamics
Description: The change in cardiac hemodynamics as measured by echocardiography. The E/e' ratio is a marker used to evaluate the left ventricular (LV) filling pressures during exercise. An E/e' ratio of <8 is considered to be normal, a ratio >15 is considered to reflect an increase in the LV filling pressure.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Sodium Nitrite
Number analyzed (Participants) | 16 | 16
ratio | 1.1 (3.2) | -0.2 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite; Test type: Superiority; p = 0.538, t-test, 2 sided

4. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self-administered questionnaire that provides a measure of symptoms and physical limitations associated with heart failure. The overall summary score ranges from 0-100, where the higher the score the better the health status.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Sodium Nitrite
Number analyzed (Participants) | 36 | 36
score on a scale | 6.1 (12.2) | 4.9 (14.1)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite; Test type: Superiority; p = 0.708, t-test, 2 sided

5. Secondary Outcome: Change in Six Minute Walk Test
Description: The six minute walk test is an exercise test used to assess aerobic capacity and endurance. The total distance covered over six minutes is measured in meters.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Sodium Nitrite
Number analyzed (Participants) | 35 | 36
meters | 31 (37) | 37 (46)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite; Test type: Superiority; p = 0.496, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the initiation of any study procedures to the end of the study treatment follow-up, approximately a total of 14 weeks for each participant.
Arm/Group | Placebo | Sodium Nitrite
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 3/36 | 7/37
Other Adverse Events (participants affected / at risk) | 36/36 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Sodium Nitrite (N=37)
Severe Chest/Neck/Jaw Pain (Cardiac disorders) | 1 (1) | 2 (2)
Serious Fall Resulting in Injury (General disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness/Lightheadedness (General disorders) | 1 (1) | 0 (0)
Shortness of Breath - Worsening Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Arrhythmia (General disorders) | 0 (0) | 1 (1)
Syncope/Stent placement (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Sodium Nitrite (N=37)
Cough (General disorders) | 7 (8) | 10 (12)
Chest pain (General disorders) | 8 (9) | 11 (14)
Dizziness (General disorders) | 14 (19) | 22 (30)
Edema (General disorders) | 1 (2) | 2 (2)
Fatigue (General disorders) | 6 (10) | 3 (3)
Upset stomach/diarrhea (Gastrointestinal disorders) | 5 (6) | 12 (16)
Headache (General disorders) | 8 (8) | 10 (10)
Cold/SoreThroat/Flu (General disorders) | 13 (14) | 13 (18)
General Minor Injury - Fall/Bruise/Cut (General disorders) | 4 (4) | 7 (8)
Miscellaneous - Blister/Bloody nose/Cataract/Dry Mouth/Acne (General disorders) | 11 (12) | 20 (29)
Nausea (General disorders) | 6 (8) | 5 (6)
Memory Loss (General disorders) | 2 (2) | 0 (0)
Numbness/Pins and Needles (General disorders) | 1 (1) | 1 (1)
Muscle and Joint Pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 15 (17)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Mood Changes - Depressed/Edgy/Forgetful (General disorders) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2)
Shortness of Breath (General disorders) | 6 (8) | 10 (14)
Bad Taste in Mouth (General disorders) | 1 (1) | 2 (2)
Weight Gain (General disorders) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Black Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening Renal Function (General disorders) | 0 (0) | 1 (1)
Revascularization (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Manufacturer discontinuation of the inhaled drug supply forced the investigator to modify the study and change the route of administration of sodium nitrite from inhaled to oral. The oral formulation achieved similar pharmacokinetics and therefore it was scientifically justified to combine the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT02713126/Prot_SAP_000.pdf